CLINICAL TRIAL: NCT04409561
Title: A Study to Establish a Reference Range for abioSCOPE® Device With the PSP Assay in a Generally Healthy Adult Population
Brief Title: Reference Range for abioSCOPE® Device With the PSP Assay in a Generally Healthy Adult Population
Status: Completed | Type: Observational
Sponsor: Abionic SA (Industry)
Collaborators: Boston Biomedical Associates (Other); Ocean State Clinical Coordinating Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: AB-PSP-003
Record Dates: First submitted 2020-05-14; First posted 2020-06-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Sepsis; Septic Shock; Healthy
Keywords: Sepsis; Pancreatic Stone Protein; Immunoassay; Abionic; Healthy population; Point-of-care device
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — 9 mL K3-EDTA anticoagulated venous whole blood and 9 mL lithium heparin anticoagulated venous whole blood will be collected, processed in plasma and stored until the shipment to the sponsor for PSP measurement on the abioSCOPE device with IVD CAPSULE PSP kits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Interventions: This patient pool shall be representative of the US population in term of the relative proportion of race/ethnicities. In addition, the population shall be enriched with patients above 60 year old as the target population of the PSP test is mostly the elderly.
  Interventions: Device: Blood collection

INTERVENTIONS:
Device: Blood collection — 9 mL K3-EDTA anticoagulated venous whole blood and 9 mL lithium heparin anticoagulated venous whole blood will be collected, processed in plasma and stored until the shipment to the sponsor for PSP measurement on the abioSCOPE device with IVD CAPSULE PSP kits

SUMMARY:
This is a single center, prospective, biomarker-result-blinded observational study evaluating immunoassay measurements of pancreatic stone protein (PSP) performed on Abionic's abioSCOPE device with the PSP assay on generally healthy adults representative of the US population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years.
2. Apparently healthy as determined by a subject questionnaire.

Exclusion Criteria:

1) Current diagnosis, or history, of any underlying major medical condition determined by the investigator, including but not limited to:

1. Heart disease
2. Stroke
3. Renal disease
4. Liver disease
5. Pancreatic disease
6. Chronic obstructive pulmonary disorder
7. Bleeding disorders
8. Hypercalcitoninemia
9. HIV AIDS
10. Receiving antibiotic therapy
11. Suspected infection
12. Immunosuppression

    2) Underwent procedures related to sepsis, or diagnosed with sepsis, within the last 12 months.

    3) Current diagnosis of uncontrolled hypertension, hypotension, or diabetes.

    4) Diagnosis of bacterial, fungal, or malaria infection within the last 3 months that required antimicrobial treatment.

    5 )Experienced severe trauma, surgery, cardiac shock, or severe burn within the previous 3 months requiring medical care.

    6) Current diagnosis of cancer within the last 12 months.

    7) Received immunotherapy to stimulate or inhibit cytokines within the last 12 months.

    8) Hospitalization for more than 24 hours within the last 3 months.

    9) Reported as currently pregnant or nursing a child

    10) Unable or unwilling to provide the required blood sample for testing.

    11) Any other criteria that, in the opinion of the investigator, would render the participant unsuitable for inclusion in the trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 150 generally healthy adults. This patient pool shall be representative of the US population in term of the relative proportion of race/ethnicities. In addition, the population shall be enriched with patients above 60 year old as the target population of the PSP test is mostly the elderly.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Determination of reference range interval of PSP | Day 1
  To determine the reference range intervals of PSP values measured using abioSCOPE device with the PSP assay in a generally healthy population representative of the US population.

SECONDARY OUTCOMES:
Collect medical data of healthy volunteer | Day 1
  To collect medical data from the 150 study participants using a volunteer questionnaire
Obtain well characterised samples library to be used for future tests development | Day 1
  Whole blood collection from 150 healthy subject to be used for future tests development.

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Health St. Vincent, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided